CLINICAL TRIAL: NCT00358085
Title: Expertise Based Randomized Controlled Trial of Open Versus Endovascular Repair of Abdominal Aortic Aneurysms: A Pilot Study
Brief Title: NExT ERA: National Expertise Based Trial of Elective Repair of Abdominal Aortic Aneurysms: A Pilot Study
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other)
Organization: McMaster University (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Record Dates: First submitted 2006-07-26; First posted 2006-07-28 (Estimated); Last update posted 2006-07-28 (Estimated); Status verified 2006-07

CONDITIONS: Aortic Aneurysm, Abdominal
Keywords: Endovascular; Vascular Surgical Procedures; Aneurysm; Expertise Based Methodology
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Aneurysm

INTERVENTIONS:
Procedure: Endovascular Repair of Abdominal Aortic Aneurysm
Procedure: Conventional open repair of Abdominal Aortic Aneurysm

SUMMARY:
Objectives.

To study the feasibility of an expertise-based randomized controlled trial (RCT) testing the role of traditional surgery (OPEN) versus endovascular repair (EVAR) for abdominal aortic aneurysms (AAA).

Study design.

We will conduct an expertise-based RCT comparing OPEN to EVAR of non-urgent abdominal aortic aneurysms in patients referred to vascular surgeons practicing at Hamilton Health Sciences, to determine the rate of death and other complications. Quality of life and status at 6 months will also be recorded. The ultimate goal is to determine the feasibility of conducting a pragmatic expertise-based RCT and to inform a future larger study at a national level.

DETAILED DESCRIPTION:
Background. The prevalence in individuals over 65 years of age is 6% (95% Confidence Interval [CI] 5 - 6)(1-4)in men and 1% (95% CI 1 - 2) in women.(5) AAA confers a risk of spontaneous rupture and death: the in-hospital mortality rate of ruptured aneurysms in Ontario was estimated at 40.8%.(6) Prevention of spontaneous rupture is the rationale for surgical intervention. Evidence has established that elective open surgery for AAAs > 5.5cm increases survival(7), but the 30-day perioperative mortality for elective open repair of AAA can be as high as 8%.(8-17) Phase I and II trials have found that endovascular repair is a 'viable and effective treatment' for AAA disease (18;19); the theoretical benefits include avoidance of laparotomy and no aortic clamping.

The results of RCTs (DREAM and EVAR-1)(20;21) have left unanswered the indications for endovascular repair compared with open surgery because of problems with definition of outcomes, lack of statistical power, and surgical expertise (surgeons needed to have done at least 20 surgeries with or without supervision). The only studies addressing the issue of expertise in this field suggests that 60 EVAR need to be done to achieve less than 10% complications (22), and a time interval of less than 10 days between procedures is important to maintain competence and reduce complications.(23) In addition the two RCTs used a conventional design and we have reported that this has intrinsic pitfalls. We argued that in surgery, particularly when a new technique is studied, another approach should be used: the expertise based RCT.(24) Conventional RCTs typically randomize participants to one of two interventions (A or B) and the same clinician give intervention A to some participants and B to others. The expertise based randomized controlled trial, randomizes participants to clinicians with expertise in intervention A or clinicians with expertise in intervention B, and the clinicians perform only the procedure for which they have expertise.

Study Design/Participants

We will conduct an expertise based RCT comparing open repair with EVAR repair of elective infrarenal AAAs. This is a pilot to determine the feasibility of a large pragmatic expertise based RCT of open versus EVAR repair.

We will consider all patients with an AAA determined to require non-urgent repair after assessment by one of the participating surgeons. The second inclusion criterion is that the blinded measurement team must deem a patient to fulfill the anatomic eligibility criteria.

Location of Investigation

This pilot study will be conducted at a single institution: Hamilton Health Sciences, Hamilton General Hospital. This centre will serve as the coordinating site for the future multicentre randomized controlled trial, and based on the high volume practices of the surgeons at the Hamilton General Hospital, will likely provide the largest pool of eligible patients. Protocols and standard operating procedures for a single site will be developed for this pilot, which will become standards for the larger trial. The decision to use a single centre for this pilot study is based in the high expected surgical volume that makes our recruitment rate realistic, in addition to the cost savings of conducting a trial close to investigators and surrounded by known infrastructure.

Patient Recruitment

Once a patient is deemed eligible, the study nurse will provide the patient with details of the study protocol and explanation of goals of the investigation, and obtain informed consent.

Randomization and Allocation

The study nurse will be contacted by the surgeons' offices to screen all patients referred to participating vascular surgeons on the first visit to the office and submit a standardized electronic form accessible on a secure, encrypted website. This will document baseline demographics for referred patients including key eligibility criteria. If these are met, the study nurse will contact the patient, explain the study, determine the remaining eligibility criteria and obtain consent. The nurse will use the electronic database to randomly allocate the patient to open or endovascular repair. We will ensure concealment of allocation through the use of a randomization and allocation process housed on an encrypted website monitored by a data coordinator external to the study protocol. This process has been successfully developed within the St Joseph's Nephrology, Thromboembolism and Vascular research group. Randomization using random-sized permuted block technique will ensure balanced distribution of patients and concealment of allocation. Once allocation has occurred, the study nurse will coordinate patient appointments to the appropriate surgeon. Patients who do not meet eligibility requirements will return to their original surgeon for disclosure of results and treatment.

Patient Follow-up

The study nurse will meet the patient, document baseline characteristics and perform blood work at the preoperative clinic visit. The study nurse will see patients daily after surgery, arrange daily blood work and document all outcome events using standardized case report forms until discharged from hospital. An outcome assessor committee independent of the study and blinded to treatment allocation will adjudicate all outcome events. The study nurse will see all patients at 3-month intervals for 6 months. The use of a 6-month outcome threshold is for purposes of assessing feasibility in this pilot study only. The larger multicentre trial will plan to evaluate outcomes up to five years, addressing the long term concerns that have been raised in RCTs.

Evaluation of Pilot Objectives

We will consider the pilot study a success if we can:

1. Recruit 30 patients in 40 weeks
2. Obtain a complete follow-up on 95% of the trial patients
3. Demonstrate the feasibility of using a web-based system to randomize and follow patients in this trial, and for outcome adjudication, and
4. Document the resources (e.g., personnel time) required to conduct this trial.

Ethical Considerations

All patients in this study will provide informed consent prior to participation, and the protocol will be reviewed by the Ethics Review Board of Hamilton Health Sciences.

Reference List

1. Lindholt JS, Juul S, Fasting H, Henneberg EW. Screening for abdominal aortic aneurysms: single centre randomised controlled trial. BMJ, 330: 750.
2. Ashton HA, Buxton MJ, Day NE et al. The Multicentre Aneurysm Screening Study (MASS) into the effect of abdominal aortic aneurysm screening on mortality in men: a randomised controlled trial. Lancet, 360: 1531-1539.
3. Norman PE, Jamrozik K, Lawrence-Brown MM et al. Population based randomised controlled trial on impact of screening on mortality from abdominal aortic aneurysm. BMJ, 329: 1259.
4. Scott RA, Vardulaki KA, Walker NM, Day NE, Duffy SW, Ashton HA. The long-term benefits of a single scan for abdominal aortic aneurysm (AAA) at age 65. European Journal of Vascular & Endovascular Surgery, 21: 535-540.
5. Scott RA, Bridgewater SG, Ashton HA. Randomized clinical trial of screening for abdominal aortic aneurysm in women. Br.J.Surg., 89: 283-285.
6. Dueck AD, Kucey DS, Johnston KW, Alter D, Laupacis A. Survival after ruptured abdominal aortic aneurysm: effect of patient, surgeon, and hospital factors. J.Vasc.Surg., 39: 1253-1260.
7. Mortality results for randomised controlled trial of early elective surgery or ultrasonographic surveillance for small abdominal aortic aneurysms. The UK Small Aneurysm Trial Participants. Lancet, 352: 1649-1655.
8. Ernst CB. Abdominal aortic aneurysm. N.Engl.J.Med., 328: 1167-1172.
9. Zarins CK, Harris EJ, Jr. Operative repair for aortic aneurysms: the gold standard. J.Endovasc.Surg., 4: 232-241.
10. Lawrence PF, Gazak C, Bhirangi L et al. The epidemiology of surgically repaired aneurysms in the United States. J.Vasc.Surg., 30: 632-640.
11. Heller JA, Weinberg A, Arons R et al. Two decades of abdominal aortic aneurysm repair: have we made any progress? J.Vasc.Surg., 32: 1091-1100.
12. Galland RB. Mortality following elective infrarenal aortic reconstruction: a Joint Vascular Research Group study. Br.J.Surg., 85: 633-636.
13. Johnston KW, Scobie TK. Multicenter prospective study of nonruptured abdominal aortic aneurysms. I. Population and operative management. J.Vasc.Surg., 7: 69-81.
14. Bradbury AW, Adam DJ, Makhdoomi KR et al. A 21-year experience of abdominal aortic aneurysm operations in Edinburgh. Br.J.Surg., 85: 645-647.
15. Bayly PJ, Matthews JN, Dobson PM, Price ML, Thomas DG. In-hospital mortality from abdominal aortic surgery in Great Britain and Ireland: Vascular Anaesthesia Society audit. Br.J.Surg., 88: 687-692.
16. Huber TS, Wang JG, Derrow AE et al. Experience in the United States with intact abdominal aortic aneurysm repair. J.Vasc.Surg., 33: 304-310.
17. Kazmers A, Jacobs L, Perkins A, Lindenauer SM, Bates E. Abdominal aortic aneurysm repair in Veterans Affairs medical centers. J.Vasc.Surg., 23: 191-200.
18. Thomas SM, Gaines PA, Beard JD. Short-term (30-day) outcome of endovascular treatment of abdominal aortic aneurism: results from the prospective Registry of Endovascular Treatment of Abdominal Aortic Aneurism (RETA). Eur.J.Vasc.Endovasc.Surg., 21: 57-64.
19. Harris PL, Buth J, Mialhe C, Myhre HO, Norgren L. The need for clinical trials of endovascular abdominal aortic aneurysm stent-graft repair: The EUROSTAR Project. EUROpean collaborators on Stent-graft Techniques for abdominal aortic Aneurysm Repair. J.Endovasc.Surg., 4: 72-77.
20. Prinssen M, Verhoeven EL, Buth J et al. A randomized trial comparing conventional and endovascular repair of abdominal aortic aneurysms. N.Engl.J.Med., 351: 1607-1618.
21. Greenhalgh RM, Brown LC, Kwong GP, Powell JT, Thompson SG. Comparison of endovascular aneurysm repair with open repair in patients with abdominal aortic aneurysm (EVAR trial 1), 30-day operative mortality results: randomised controlled trial. Lancet, 364: 843-848.
22. Forbes TL, DeRose G, Kribs SW, Harris KA. Cumulative sum failure analysis of the learning curve with endovascular abdominal aortic aneurysm repair. J.Vasc.Surg., 39: 102-108.
23. Lobato AC, Rodriguez-Lopez J, Diethrich EB. Learning curve for endovascular abdominal aortic aneurysm repair: evaluation of a 277-patient single-center experience. J.Endovasc.Ther., 9: 262-268.
24. Devereaux PJ, Bhandari M, Clarke M et al. Need for expertise based randomised controlled trials. BMJ, 330: 88.

ELIGIBILITY:
Inclusion Criteria:

All patients with an AAA determined to require non-urgent repair after assessment by one of the participating surgeons will be considered. Patients must meet two eligibility criteria: Medical and Anatomic.

Medical Fitness for surgery will mean that the patient is a candidate for elective open repair, and has none of the exclusion criteria listed below.

Anatomic Eligibility will be judged by the endovascular measurement team, and will be based on a score of < 3 on the following scale. (This scale was developed at our centre and is currently being validated.)

1. Neck Length (20 - 15 mm = 1; 14 - 10 mm = 2)
2. Quality of Neck (Thrombus 90 -180 º = 1, 181-270 º = 2; calcification 90 -180 º = 1; 181-270 º = 2)
3. Presence/absence side branches (IMA or lumbar vessels = 1; IMA and lumbar vessels or other = 2)
4. Landing zone (aneurysmal or occlusive disease = 1; aneurysmal and occlusive disease = 2;
5. Degree of calcification of aorta (25 - 50% calcification = 1; > 50% = 2)
6. Access (stenosis = 1; stenosis and tortuosity =2)
7. Stenting of accessory renal arteries necessary
8. Embolization of internal iliac artery necessary

Definition of Surgical Experts

Expertise in endovascular surgery will be determined by completion of a vascular residency at a credentialed academic centre, a period of study in a formal training programme dedicated to acquiring endovascular expertise, and experience with at least 60 previous EVAR procedures.30

Expertise in open aortic repair will require completion of an accredited vascular surgery residency programme and demonstration of expertise by having completed at least 100 consecutive elective AAA repairs in their career.32

Endovascular Measurement Team The Endovascular Measurement team consists of at least one vascular surgeon with expertise in endovascular surgery, at least one vascular fellow in his/her first or second year of training and a representative from an endovascular graft specialist who is familiar with graft measurement and deployment. This team, blinded to patient demographics and surgical fitness, will judge anatomic eligibility.

Exclusion Criteria:

1. Exclusion due to Medical Risk: Patients with severe cardiac or respiratory disease that limits their activities of daily living and would make them ineligible for open repair. BMI greater than 45. Any known diagnosis or condition that renders a lift span of less than 2 years based on available and tolerable treatments.
2. Exclusion due to Aneurysm Factors: Patients with ruptured or symptomatic aneurysms requiring urgent surgery. Any aneurysm that extends proximal to the renal arteries (suprarenal), involves the renal arteries or is less than 15mm distal to the level of the lowest renal artery.
3. Exclusion due to Operative Factors: Patients with multiple previous laparotomies making open repair contraindicated due to adhesions (a 'hostile abdomen'). Any patients with stomas or exteriorized bowel. Patients with previous abdominal radiation, Fitz-Hugh-Curtis, or history of other conditions that would render open operative intervention contraindicated.

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30
Dates: Start 2006-09; Study Completion 2008-01

PRIMARY OUTCOMES:
Mortality from the time of randomization until hospital discharge or 30-days after surgery

SECONDARY OUTCOMES:
Non-fatal myocardial infarction.
End organ ischemic event rates (including Renal Failure, Limb ischemia, Bowel ischemia, Non-fatal stroke)
Reintervention
Quality of life
Success of repair
Mortality at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Tara M Mastracci, MD, FRCSC, Principal Investigator — McMaster University; Claudio S Cina, MD, Spec Chir(It), FRCSC, MSc, Study Director — McMaster University; Catherine M Clase, MD, FRCSC, MSc, Study Director — McMaster University; PJ Devereaux, MD, FRCSC, PhD, Study Director — McMaster University
Locations (1):
- McMaster University, Hamilton General Hospital, Hamilton, Ontario, Canada